CLINICAL TRIAL: NCT04701632
Title: Prevalence and Variables Associated With Depression in Subjects With Chronic Wounds Using PHQ-9 as a Screening Tool
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 055.WCHC.2019.D
Record Dates: First submitted 2019-11-04; First posted 2021-01-08 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study is to complete a retrospective chart review of subjects who were treated at the Wound Care Clinic at Methodist Dallas Medical Center, presented for treatment between June 2018 and February 2019, and were administered the PHQ-9. The study aims to measure the prevalence of depression in this sample, feasibility of using PHQ-9 in this patient population, and identifying variables and functional impairment associated with clinically significant depression.

DETAILED DESCRIPTION:
The study will review medical records of new patients who presented to the Wound Care Center at Methodist Dallas Medical Center between June 2018 and February 2019. These patients were all administered PHQ-9 as part of a quality improvement project. The medical records included for analysis will be from male and female patients aged 18 years or older. The medical records will be reviewed for the following information: general demographics, information including age, sex, ethnicity, race, PHQ-9 score (total and individual items), medical conditions, wound history, past medical history, general symptoms, abuse and suicide risk, activities of daily living, motivation assessment, mental status, and pain ratings. This information will be used to measure the prevalence of clinically significant depression in the sample, which is the primary aim. We will also use the data to establish factors and variables correlated with the presence and severity of clinically significant depression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Received care at the Wound Care Center at Methodist Dallas Medical Center between June 2018 and February 2019
3. Completed a PHQ-9 form at the time of initial evaluation/examination

Exclusion Criteria:

1. Patients less than 18 years of age will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: new patients who presented to the Wound Care Center at Methodist Dallas Medical Center between June 2018 and February 2019.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2022-11-14 (Estimated); Study Completion 2022-11-14 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 score | Through study completion, an average of 1 year
  to measure the prevalence of clinically significant depression defined as a PHQ-9 score of equal to or greater than 10.

CONTACTS AND LOCATIONS:
Overall Officials: Asma Khatoon, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Wound care & Hyperbaric Clinic, Dallas, Texas, United States